CLINICAL TRIAL: NCT01835847
Title: Tipepidine for Adolescent Depression
Brief Title: An Open Study of Tipepidine Hibenzate in Adolescent Patients With Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Tsuyoshi Sasaki, Assistant Professor, Chiba University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G24062
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Depression; Adolescent
MeSH Terms: conditions — Depression | interventions — tipepidine

ARMS (1):
- A single-arm study (Experimental)
  Interventions: Drug: Tipepidine Hibenzate

INTERVENTIONS:
Drug: Tipepidine Hibenzate

SUMMARY:
Accumulating evidence suggests a role of G protein-coupled inwardly-rectifying potassium (GIRK) channel in the pathology of excitement of nerve, and the medicine with the action (like the Tipepidine Hibenzate) is expected as a new curative medicine of adolescent depression.

The purpose of this research is to confirm the effect by carrying out the additional dosage of the Tipepidine Hibenzate to the adolescent patients with depression.

If suggestion is obtained by this research about the effect on adolescent patients with depression of Tipepidine Hibenzate, it can contribute to development of the medical treatment of adolescent patients with depression.

ELIGIBILITY:
[Inclusion Criteria]

1. Depressive Episode for ICD-10 criteria.
2. Patients are treated with antidepressants (SSRI ; Fluvoxamine, Paroxetine, Sertraline, Escitalopram, SNRI ; Milnacipran, Duloxetine, NaSSa; Mirtazapine), mood stabilizers (Lithium, Sodium Valproate, Carbamazepine, Lamotrigine), atypical antipsychotics (Risperidone, Olanzapine, Quetiapine, Perospirone, Aripiprazole, Blonanserin, Paliperidone) or not treated.
3. Patients are stable for 4-weeks for medication.

[Exclusion Criteria]

1. Patients with a previous hypersensitivity to Tipepidine Hibenzate.
2. Patients treated with typical antipsychotics and antidepressants except inclusion criteria 2. and mood stabilizers except inclusion criteria 2.
3. Pregnant or breast-feeding women

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Children's Depression Rating Scale, Revised (CDRS-R) | Changes from baseline in CDRS-R at 4-weeks
  The CDRS-R is a brief rating scale based on a semi-structured interview with the child (or an adult informant who knows the child well). Designed for 6- to 12-year-olds, and successfully used with adolescents, it can be administered in just 15 to 20 minutes and easily scored in a few minutes more. The interviewer rates 17 symptom areas (including those that serve as DSM-IV criteria for a diagnosis of depression):

SECONDARY OUTCOMES:
Depression Self-Rating Scale for Children (DSRS-C) Japenese Version | Changes from baseline in DSRS-C at 4-weeks
  DSRS-C is easy to use and has a predictive value comparable with that of a psychiatric global rating of depressed appearance and history of depression obtained at interview. There was confirmation that the DSRS-C can tap an internal dimension of depression and that children are able to evaluate their feeling states.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Chiba University School of Medicine, Chiba, Chuo-ku, Japan

REFERENCES:
- [Result] Sasaki T, Hashimoto K, Tachibana M, Kurata T, Kimura H, Komatsu H, Ishikawa M, Hasegawa T, Shiina A, Hashimoto T, Kanahara N, Shiraishi T, Iyo M. Tipepidine in adolescent patients with depression: a 4 week, open-label, preliminary study. Neuropsychiatr Dis Treat. 2014 May 5;10:719-22. doi: 10.2147/NDT.S63075. eCollection 2014. No abstract available. PMID 24833905